CLINICAL TRIAL: NCT00781482
Title: Positron Emission Tomography Assessment of the Central Nervous System Effects of Eszopiclone and Zolpidem
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Sponsor elected not to conduct study at this time.
Sponsor: Kettering Health Network (Other)
Collaborators: Abiant, Inc. (Industry); Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Joseph Mantil, MD, PhD, Kettering Health Network
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 07-104-SEPR
Record Dates: First submitted 2008-10-27; First posted 2008-10-29 (Estimated); Last update posted 2016-02-26 (Estimated); Status verified 2016-02

CONDITIONS: Healthy
Keywords: Positron Emission Tomography; GABA receptor binding; Hypnotic Drugs; Eszopiclone; Zolpidem; [11-C] Flumazenil; Molecular imaging of the brain
MeSH Terms: interventions — Eszopiclone; Zolpidem

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): This is a crossover study. Each study drug will be administered (one at a time and in random order) to each subject on separate occasions over the course of the study.
  Interventions: Drug: eszopiclone, zolpidem, placebo

INTERVENTIONS:
Drug: eszopiclone, zolpidem, placebo — In random order, each subject will receive one study drug per visit over three visits. Visits will occur about 1 week apart. Each subject will eventually receive eszopiclone 3 mg., zolpidem 10 mg., and a placebo. PET scans will be done 1-2 hours after each dose.
  Other Names: Lunesta; Ambien

SUMMARY:
This study will compare the interactions of a placebo and two FDA-approved sleeping medications, Eszopiclone (Lunesta) and Zolpidem (Ambien), with certain chemical receptors in the brain. We want to show that we can use positron emission tomography images to measure the binding of these medications to the receptors.

DETAILED DESCRIPTION:
We will enroll 4 normal, healthy, adult male volunteers who will undergo screening tests (labs, EKGs, medical history, physical exam, and MRI of the brain) for safety. If eligible, they will return for three separate positron emission tomography (PET) scans. Over the course of the three study visits, each subject will receive eszopiclone (Lunesta), zolpidem (ambien) and a placebo in random order.

After each medication or placebo dose, a PET scan will be done using a [11-C] flumazenil (Romazicon). The flumazenil will help us measure the binding of the study medications to chemical receptors called GABA receptors in certain parts of the brain.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Males age 18 to 35 inclusive
* Body Mass Index 18 to 30
* Willing to adhere to prohibitions and restrictions specified in protocol
* Must give informed consent.

Exclusion Criteria:

* Clinically significant abnormal lab values for chemistry, hematology or urinalysis at screening.
* Clinically significant abnormal physical exam, vital signs, or 12-lead EKG at screening
* Significant history of or current significant medical illness.
* Significant history of or current psychiatric or neurological illness or sleep apnea.
* Participation in another research study involving exposure to ionizing radiation within the last 12 months.
* Any clinically significant MR abnormality which may be relevant to the study.
* Metal implants which are relevant for MR or PET procedures or data.
* History of epilepsy or fits or unexplained blackouts.
* Serology positive for Hepatitis B surface antigen, Hepatitis C antibodies, or HIV antibodies.
* Positive urine screen for drugs of abuse.
* Positive alcohol screen.
* Known or suspected alcoholism or drug addiction even if currently abstaining
* Drinks on average more than 8 cups of coffee, tea, cocoa, or cola per day.
* Smoking cigarettes within 3 months prior to study drug administration.
* Clinically significant acute illnes within 7 days of study drug administration.
* Claustrophobia.
* Donation of 1 or more units of blood (approximately 450ml), or acute loss of an equivalent amount of blood within 90 days prior to study drug administration.
* Have received an experimental drug or used an experimental medical device within 90 days of planned start of treatment with drugs for this study.
* Use of any prescription or over the counter medication, or herbal medication (not including non-steroidal anti-inflammatory drugs) within 2 weeks of the first PET scan. Of particular concern would be GABA-ergic compounds and CYP3A4 inhibitors. Exclusion should also be considered if the subject has taken a drug with a long half-life (or of any metabolite) even if taken outside the two week time window. However, the subject can still be enrolled if, in the opinion of the investigator, such medication taken in that timeframe will not interfere with the results of the study.
* Psychological or emotional problems that would render the informed consent invalid or limit the ability of the subject to comply with the study requirements.
* Any condition that in the opinion of the investigator would complicate or compromise the study, or the well-being of the subject.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
We will measure GABA receptor binding by PET imageing after each dose of study medication or placebo. | PET scans will occur within 1-2 hours after study drug or placebo administration. Visits will occur approximately 1 week apart. . Subjects will have visits scheduled over approximately 6 weeks, including screening, scanning visits, and follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph C Mantil, MD, PhD, Principal Investigator — Kettering Health Network
Locations (1):
- Kettering Medical Center, Kettering, Ohio, United States